CLINICAL TRIAL: NCT04872998
Title: Vascular Dysfunction During Physical Inactivity: Role of Oxidative Stress
Brief Title: Vascular Dysfunction During Physical Inactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Joel Trinity, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #111321; UL1TR002538 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2021-08

CONDITIONS: Aging; Vascular Endothelium; Skeletal Muscle
Keywords: Reduced Activity; Muscular Atrophy; Vascular Dysfunction
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Activity (Experimental): Reduction of daily step count by 70% for two weeks, followed by two week recovery to normal activity level
  Interventions: Behavioral: Step Count Reduction

INTERVENTIONS:
Behavioral: Step Count Reduction — Subjects reduce daily step counts by approximately 70% through monitoring and recording from step-count monitor

SUMMARY:
Prolonged periods of reduced activity are associated with decreased vascular function and muscle atrophy. Physical inactivity due to a sedentary lifestyle or acute hospitalization is also associated with impaired recovery, hospital readmission, and increased mortality. Older adults are a particularly vulnerable population as functional (vascular and skeletal muscle mitochondrial dysfunction) and structural deficits (loss in muscle mass leading to a reduction in strength) are a consequence of the aging process. The combination of inactivity and aging poses an added health threat to these individuals by accelerating the negative impact on vascular and skeletal muscle function and dysfunction. The underlying factors leading to vascular and skeletal muscle dysfunction are unknown, but have been linked to increases in oxidative stress. Additionally, there is a lack of understanding of how vascular function is impacted by inactivity in humans and how these changes are related to skeletal muscle function. It is the goal of this study to investigate the mechanisms that contribute to disuse muscle atrophy and vascular dysfunction in order to diminish their negative impact, and preserve vascular and skeletal muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have recently undergone surgery or injury requiring inactivity

Exclusion Criteria:

* Cardiac abnormalities considered exclusionary by the study physician (congestive heart failure, coronary artery disease, right-to-left shunt)
* Uncontrolled endocrine or metabolic disease
* Glomerular filtration rate < 45 mL/min/1.73 m^2 or evidence of kidney disease or failure
* Vascular disease or risk factors of peripheral atherosclerosis
* Risk of deep vein thrombosis including family history of thrombophilia, pulmonary emboli, deep vein thrombosis
* Use of anticoagulant therapy
* Elevated systolic pressure > 180 or a diastolic blood pressure > 110
* Implanted electronic devices such as pacemakers, infusion pumps, stimulators
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Currently on a weight-loss diet or body mass index > 35 kg/m^2
* Inability to abstain from smoking for duration of study
* History of > 20 pack per year smoking
* Positive for human immunodeficiency virus, hepatitis B or hepatitis C
* Recent anabolic or corticosteroids use (within 3 months)
* Subjects with hemoglobin or hematocrit lower than accepted lab values
* Agitation/aggression disorder
* History of stroke with motor disability
* Recent history (< 12 months) of gastrointestinal bleed
* Depression diagnosis
* Alcohol or drug abuse
* Liver disease (AST/ALT 2 times above the normal limit, hyperbilirubinemia)
* Respiratory disease (acute upper respiratory infection, history of chronic lung disease with resting oxygen saturation < 97% on room air)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Trinity, Ph.D., Principal Investigator — University of Utah
Locations (1):
- VA Medical Center Building, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Activity: Reduction of daily step count by 70% for two weeks
  Step Count Reduction: Subjects reduce daily step counts by approximately 70% through monitoring and recording from step-count monitor
Period: Overall Study
Arm/Group | Reduced Activity
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Activity
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Vascular Function
Description: The flow rate of brachial artery measured by flow-mediated dilation (FDM). Doppler ultrasound will be used to determine brachial artery vascular function. Specifically, this assessment will include the measurement of flow rate and artery diameter at rest and in response to flow mediated dilation.
Time Frame: Baseline, during reduced activity (2 weeks) and 2 weeks post reduced activity (4 weeks)
Measure: Mean (Standard Deviation); unit: percent vasodilation
Arm/Group | Reduced Activity
Number analyzed (Participants) | 14
percent vasodilation
  Baseline FMD | 5.1 (5.1)
  During reduced activity | 3.1 (2.4)
  2 week post reduced activity | 4.4 (3.4)

2. Secondary Outcome: Popliteal Artery Vascular Function
Description: Flow rate of popliteal artery measured by flow-mediated dilation (FMD). Doppler ultrasound will be used to determine popliteal artery vascular function. Specifically, this assessment will include the measurement of flow rate and artery diameter at rest and in response to flow mediated dilation.
Time Frame: Baseline, during reduced activity (2 weeks) and 2 weeks post reduced activity (4 weeks)
Measure: Mean (Standard Deviation); unit: percent vasodilation
Arm/Group | Reduced Activity
Number analyzed (Participants) | 14
percent vasodilation
  Baseline FMD | 4.5 (4.5)
  During reduced activity | 2.4 (2.1)
  2 weeks post reduced activity | 3.6 (2.3)

3. Secondary Outcome: Leg Microvascular Function
Description: Flow rate of leg microvasculature assessed by passive leg movement (PLM). Doppler ultrasound will be used to determine leg microvasculature function. Specifically, this assessment will include the measurement of flow rate at rest and in response to movement.
Time Frame: Baseline, during reduced activity (2 weeks) and 2 weeks post reduced activity (4 weeks)
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Reduced Activity
Number analyzed (Participants) | 14
ml/min
  Baseline FMD | 385 (313)
  During reduced activity | 311 (202)
  2 weeks post reduced activity | 412 (290)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Reduced Activity
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04872998/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT04872998/ICF_001.pdf